CLINICAL TRIAL: NCT04229316
Title: Safety And Efficacy Assessment of the zLock Facet Fusion System- A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZygoFix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMS-3343
Record Dates: First submitted 2020-01-08; First posted 2020-01-18 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-02

CONDITIONS: Low Back Pain
Keywords: stabilization, facet arthritis, spondylolisthesis, stenosis
MeSH Terms: conditions — Low Back Pain; Spondylolisthesis; Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- zLock Facet Locking Implant System (Experimental)
  Interventions: Device: zLOCK Facet Stabilization System

INTERVENTIONS:
Device: zLOCK Facet Stabilization System — zLOCK Facet Stabilization System is a device intended to provide posterior stability in lumbar spine in order to reduce lumbar back pains

SUMMARY:
ZygoFix has developed a system consisting of zLOCK Facet Fusion System. The zLOCK Facet Fusion System is intended for single level stabilization of a spinal motion segment to promote bonny fusion of the joint. The system is designed for percutaneous deployment. The zLOCK implant is designed to be deployed in the facet joint thereby utilizing the body's natural mechanical structure without adding an external scaffold (see figure below).

The zLOCK implant is inserted into the facet joint space while it adapts to the joint's changing geometry. Stabilization is achieved by firm grip of each joint bone and resisting to any relative motion. The zLOCK implant is placed percutaneously and requires only one incision per side, thereby reducing the invasiveness, procedure duration and shorten the recovery period.

This pilot study was designed in order to assess the safety and effectiveness of the zLOCK system.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is scheduled for spine surgery with at least one of the following:

   When used in adjunct to an intervertebral front cage:
   * Degenerative Spondylolisthesis up to grade 2
   * Mild to Moderate Degenerative disc disease (DDD)
   * Degeneration of the facets - following validating the pain source by facet injection.

   When used stand-alone:
   * Degenerative Spondylolisthesis grade 1-2
   * Moderate to severe Stenosis with listhesis
   * Moderate to severe stenosis without listhesis (in cases that the investigator determines stabilization is required).
   * Degeneration of the facets- following validating the pain source by facet injection.
2. Claudication due to moderate to severe stenosis (central/ foraminal) as verified by imaging.
3. 18< Age < 75
4. Weight < 100Kg
5. Signed informed consent form
6. At least 3 months of unsuccessful conventional treatments

Exclusion Criteria:

1. Fusion procedure performed or required in more than one inter-vertebrae space.
2. Active systemic infection or infection localized to the site of the proposed implantation are contraindications to implantation.
3. Osteoporosis
4. Absence of posterior spinal elements including the pedicle, pars interarticularis, facet joints, spinous process and the majority of the lamina which make it unstable or not possible to place.
5. Any entity or conditions that totally preclude the possibility of fusion, i.e., cancer, kidney dialysis, or osteopenia, are relative contraindications.
6. Obesity (BMI ≥30)
7. Foreign body sensitivity
8. Alcoholism, or drug abuse
9. Subject with a cardiac pacemaker or other implanted electro medical device
10. Subject with known condition of drug abuse and/or alcoholism
11. Women who are either pregnant or nursing at the time of screening (to be verified by test in case of woman of child-bearing potential that do not practice medically acceptable methods of contraception)
12. Concurrent participation in another clinical trial using any investigational drug or device.
13. Mental disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Safety assessment - no device related reoperation | 3 months
  The safety of the zLOCK Facet Implant System will be established based on the absence of device related reoperations.

SECONDARY OUTCOMES:
Efficacy assessment - achieving facet fusion 12 months post procedure | 12 months
  The efficacy of using the zLOCK System will be determined by achieving facet fusion 12 months post procedure.
  Patient is defined "success" if facet fusion is achieved at 12 months post procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Levy, Dr, Study Director — ZygoFix
Locations (1):
- Pecs University Hospital, Pécs, Hungary